CLINICAL TRIAL: NCT00547300
Title: Tolerability of Nebivolol Compared With Metoprolol ER in Patients With Mild to Moderate Hypertension Taking Hydrochlorothiazide (HCTZ)
Brief Title: Study to Evaluate Symptoms in Patients Treated With Nebivolol or Metoprolol Extended-release (ER) for Hypertension
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Collaborators: Mylan Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NEB-MD-03
Record Dates: First submitted 2007-10-19; First posted 2007-10-22 (Estimated); Results first posted 2019-05-21 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-04

CONDITIONS: Hypertension
Keywords: Hypertension; Nebivolol; Beta blocker; Tolerability
MeSH Terms: conditions — Hypertension | interventions — Metoprolol; Nebivolol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Nebivolol (Experimental): Nebivolol 5 mg, 10 mg or 20 mg
  Interventions: Drug: Nebivolol
- Metoprolol ER (Active Comparator): Metoprolol ER 50 mg, 100 mg or 200 mg
  Interventions: Drug: Metoprolol ER

INTERVENTIONS:
Drug: Metoprolol ER — Metoprolol ER once daily, oral administration
  Arms: Metoprolol ER
Drug: Nebivolol — Nebivolol once daily, oral administration
  Arms: Nebivolol

SUMMARY:
The purpose of this study was to compare the tolerability of nebivolol to metoprolol ER in a general population of patients with mild to moderate hypertension receiving hydrochlorothiazide (HCTZ)

DETAILED DESCRIPTION:
This study was an 18-week study to evaluate the tolerability of nebivolol compared to metoprolol ER in outpatients with mild to moderate hypertension taking HCTZ. It is a multi-center, randomized, double blind (DB), active-control, parallel-group study, starting with a 4-week HCTZ run-in phase, followed by a 12-week DB treatment phase. Patients meeting the entry criteria at the end of run-in are randomized to one of two treatment groups, nebivolol or metoprolol ER. Up-titration of dose of study drug will occur if needed during the first 4 weeks of the DB phase, after which there is an 8-week stable-dose period of treatment. A 2-week double-blind withdrawal phase follows, during which tapering off study drug occurs.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ambulatory outpatients
* History of hypertension being treated with two medications, one of which must be HCTZ and the other of which must not be a beta-blocker or clonidine
* SBP of 135-155 mm Hg and/or DBP of >85 mm Hg at screening (Visit 1)
* SBP of 140-165 mm Hg and DBP > 90 mmHg at randomization (Visit 3)

Exclusion Criteria:

* Treatment with a beta-blocker or clonidine within 6 months of screening (Visit 1)
* Clinically significant respiratory disease (e.g., bronchial asthma, reactive airways disease, chronic obstructive pulmonary disease)
* Coronary artery disease requiring treatment with a calcium channel blocker or nitrates
* Clinically significant cardiovascular disease (e.g., myocardial infarction, cerebrovascular event, significant arrhythmia) within 6 months of screening (Visit 1)
* History of severe mental illness (including Major Depressive Disorder, psychosis, dementia, bipolar disorder) within 6 months of screening (Visit 1)
* Use of antipsychotic medication (e.g., dopamine receptor antagonists, serotonin dopamine receptor antagonists) or antidepressants
* Diabetes mellitus, type I or II
* Participation in a previous investigational study of nebivolol at any time
* Receipt of treatment with an investigational study drug within 30 days of screening (Visit 1)
* History of hypersensitivity to nebivolol, metoprolol ER, other beta-blockers, HCTZ, or other sulfonamide-derived drugs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2007-10-31 (Actual); Primary Completion 2008-01-02 (Actual); Study Completion 2008-01-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - Forest Research Institute 014, Birmingham, Alabama
  - Forest Research Institute 028, Beverly Hills, California
  - Forest Research Institute 054, Encinitas, California
  - Forest Research Institute 025, Roseville, California
  - Forest Research Institute 013, Tustin, California
  - Forest Research Institute 053, Vista, California
  - Forest Research Institute 052, Walnut Creek, California
  - Forest Research Institute 033, Westlake Village, California
  - Forest Research Institute 010, DeLand, Florida
  - Forest Research Institute 019, Holly Hill, Florida
  - Forest Research Institute 036, Hollywood, Florida
  - Forest Research Institute 007, Pembroke Pines, Florida
  - Forest Research Institute 009, Atlanta, Georgia
  - Forest Research Institute 006, Oxon Hill, Maryland
  - Forest Research Institute 027, Las Vegas, Nevada
  - Forest Research Institute 050, Salisbury, North Carolina
  - Forest Research Institute 039, Wilmington, North Carolina
  - Forest Investigative Site 002, Charleston, South Carolina
  - Forest Research Institute 032, Greenville, South Carolina
  - Forest Research Institute 008, Nashville, Tennessee
  - Forest Research Institute 003, Carrollton, Texas
  - Forest Research Institute 012, San Antonio, Texas
  - Forest Research Institute 048, Sugar Land, Texas
  - Forest Research Institute 040, Bountiful, Utah

REFERENCES:
- See also: Related Info — http://mylan.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient recruitment occurred over a four month period from October 2007 to January 2008 at 39 US sites.
Pre-assignment Details: All patients went through a 4 week hydrochlorothiazide (HCTZ) run-in phase before randomization.
Groups:
- Metoprolol Extended-Release (ER): Metoprolol ER 50 mg, 100 mg or 200 mg
Period: Overall Study
Arm/Group | Nebivolol | Metoprolol Extended-Release (ER)
Started | 25 | 26 (Two (2) patients were randomized in error, but no study medication taken.)
Completed | 0 (No patients completed because the study was administratively terminated.) | 0 (No patients completed because the study was administratively terminated.)
Not Completed | 25 | 26
Not completed — Study was Administratively Terminated | 25 | 24
Not completed — Did not Meet Entry Criteria | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nebivolol | Metoprolol Extended-Release (ER) | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 19 | 41
  >=65 years | 3 | 5 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (8.67) | 57.0 (9.32) | 56.0 (8.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 24
  Male | 12 | 13 | 25
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 24 | 49

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Patient Symptoms Questionnaire (PSQ) Derived Score
Description: The PSQ contained 44 possible symptoms rated from 0 (no discomfort) to 5 (extreme discomfort).
Time Frame: Measurements occured over a 14 week period, from Visit 2 (Week -2) to Visit 10 (Week 12)
Population: Formal analysis of the primary endpoint was not conducted in this abbreviated study as the study was terminated before visit 10 was reached.
Arm/Group | Nebivolol | Metoprolol Extended-Release (ER)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Peripheral Blood Pressure (BP)
Time Frame: Measurements occured over a 18 week period, from Visit 1 (Week -4) through Visit 11 (Week 14)
Population: Formal analysis of the secondary endpoint was not conducted in this abbreviated study as the study was terminated before all visits were completed. No patients completed the study.
Arm/Group | Nebivolol | Metoprolol Extended-Release (ER)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Pulse Rate
Time Frame: Measurements occured over a 18 week period, from Visit 1 (Week -4) through Visit 11 (Week 14)
Population: as for outcome 2
Arm/Group | Nebivolol | Metoprolol Extended-Release (ER)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Event data was collected over a four month period from October 2007 to January 2008.
Description: Non-serious adverse events based on the safety population of (n=49).
Arm/Group | Nebivolol | Metoprolol Extended-Release (ER)
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/26
Other Adverse Events (participants affected / at risk) | 5/25 | 3/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nebivolol (N=25) | Metoprolol Extended-Release (ER) (N=24)
Pain (General disorders) | 2 | 0
Headache (Nervous system disorders) | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1

LIMITATIONS AND CAVEATS:
Study was terminated early due to administrative reasons. Formal analyses of primary and secondary endpoints were not conducted in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor can review results communications prior to public release & can embargo communications re: results for 60 days from time submitted to sponsor for review. PI shall not disclose sponsor's confidential information. Upon sponsor's request, PI shall delete any proprietary info & shall not include raw data in the publication. On sponsor's request, PI shall delay submission for any pub while sponsor files patent applications. Any publication will give recognition to Sponsor's support.